CLINICAL TRIAL: NCT00613392
Title: Antioxidant Supplementation in Trauma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Supplement expired and unable to obtain more from company manufacturing
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-25038
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Trauma
Keywords: antioxidant; oxidant stress; trauma; free radical
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: powdered antioxidant
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: powdered cornstarch placebo

INTERVENTIONS:
Dietary Supplement: powdered antioxidant — one vial mixed with water every day orally or through enteral tube
  Arms: 1
Dietary Supplement: powdered cornstarch placebo — one vial mix with water and administer orally or via enteral tube
  Arms: 2

SUMMARY:
Administration of antioxidants to trauma patients will improve measures of oxidant stress in the blood

ELIGIBILITY:
Inclusion Criteria:

* Adult non pregnant non lactating trauma patient

Exclusion Criteria:

* GCS <6
* Renal dysfunction (cre > 2.5 mg/dl)
* Hepatic dysfunction ( TBili > 3.0 mg/dl)
* Expected survival < 48 hours
* Burns over > 20% body surface area
* Immune-deficiency syndromes
* Steroid use

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
measures of malondialdehyde level/total antioxidant status and F2 isoprostane | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Burke, MD, Study Director — Boston Medical Center